CLINICAL TRIAL: NCT01291654
Title: Paracetamol in the Treatment of Patent Ductus Arteriosus in the Premature Neonate
Brief Title: Paracetamol and Patent Ductus Arteriosus (PDA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Cathy Hammerman, Prof. Pediatrics, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SZMC-Hammerman-Acamol-2011
Record Dates: First submitted 2011-02-06; First posted 2011-02-08 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Paracetamol; Indomethacin; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Experimental): Babies with hsPDA will be treated with paracetamol 15 mg/kg/dose x 4/day for three days
  Interventions: Drug: Paracetamol
- NSAID (Experimental): Babies with hsPDA will be randomized to treatment with IV indomethacin 17 mcg/kg/hr x 36 hr
  Interventions: Drug: NSAID; Drug: D5W

INTERVENTIONS:
Drug: Paracetamol — po Paracetamol 15 mg/kg every 6 hours x 3 days
  Arms: Paracetamol
Drug: NSAID — IV indomethacin 2 mg/kg/dose for three doses at 12 hour intervals; or IV Ibuprofen 10 mg/kg infused over 15 minutes, followed by two doses of 5mg/kg each at 24 hour intervals (total of 3 doses).
  Arms: NSAID
Drug: D5W — Since the paracetamol is given q 6 hours, in order to maintain blinding of the clinical staff, a placebo (D5W) must be given intermittently between the doses of NSAID such that each infant will receive drug every 6 hours.
  Arms: NSAID

SUMMARY:
The investigators propose that paracetamol will be similarly effective to ibuprofen in treating PDA in the premature neonate, with fewer side effects.

DETAILED DESCRIPTION:
Preterm neonates with a hemodynamically significant PDA will potentially be candidates for study. After obtaining parental consent, the infants will be prospectively and randomly assigned to one of two groups: 1.po Paracetamol at a dose of 15 mg/kg every 6 hours at x 3 days or Group 2- IV indomethacin - 0.2 mg/kg/dose q 12h for three doses; or IV Ibuprofen 10 mg/kg infused over 15 minutes, followed by two doses of 5mg/kg each at 24 hour intervals (total of 3 doses).Clinical staff will be blinded as to the study group assignment of the babies and since the group 1 drug is to be given every six hours, all babies will receive a parenteral substance every 6 hours. For Group 2 infants, the intermittent doses will be IV D5W alternating with drug.All infants will fed trophic feeds (20 cc/kg/day) during the treatment for ductal closure.

ELIGIBILITY:
Inclusion Criteria:

* Echocardiographic diagnosis of hemodynamically significant patent ductus arteriosus

Exclusion Criteria:

* Major congenital anomalies
* Life-threatening infection
* Active NEC and/or intestinal perforation
* Recent (within the previous 24 hours) intraventricular hemorrhage Grade 3-4
* Urine output <1 ml per kilogram per hour during the preceding 8 hours
* Serum creatinine concentration of >1.6 mg %
* Platelet count of <60,000 per cc.

Ages: 2 Days to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Closure of the Ductus | 3 days

SECONDARY OUTCOMES:
Absence of peripheral vasoconstriction | 48 hours
  Doppler flow velocity in anterior cerebral artery, superior mesenteric artery and renal artery will be measured before and after pharmacologic treatment.
Absence of hepatotoxicity | 1 week
  Liver function will be compared between the two study groups at 1 week following completion of pharmacologic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Hebrew University Faculty of Medicine
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel